CLINICAL TRIAL: NCT06920459
Title: Zimmer Biomet Shoulder Arthroplasty Long-term Post Market Clinical Follow-up Study
Brief Title: Zimmer Biomet Shoulder Arthroplasty PMCF Study
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CMU2019-35E-EU
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Shoulder Fractures; Shoulder Arthritis Osteoarthritis; Shoulder Injury; Shoulder Pain; Degenerative Joint Disease; Arthritis Shoulder
Keywords: medical device; PMCF; Anatomic Total Shoulder Arthroplasty
MeSH Terms: conditions — Shoulder Fractures; Shoulder Injuries; Shoulder Pain; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Zimmer Biomet Total Shoulder Arthroplasty System: Patients who are having primary total shoulder arthroplasty who will receive a Zimmer Biomet Total Shoulder Arthroplasty System
  Interventions: Device: Alliance™ Glenoid

INTERVENTIONS:
Device: Alliance™ Glenoid — Total Shoulder Arthroplasty using the Alliance™ Glenoid implant

SUMMARY:
This is a multicenter, prospective, non-controlled post market surveillance study. The objectives of this study are to confirm the safety, performance, and clinical benefits of the Zimmer Biomet Shoulder Arthroplasty systems in primary anatomic shoulder arthroplasty and its instrumentation. Safety of the systems will be assessed by monitoring the frequency and incidence of adverse events. The performance and clinical benefits will be evaluated by assessment of the overall pain and functional performance, qualify of life, and radiographic parameters of all enrolled study subjects.

DETAILED DESCRIPTION:
The primary endpoint for this study will be performance assessed by improvement in the American Shoulder and Elbow Surgeons (ASES) shoulder score from baseline to 2 years (as evaluated using the overall cohort mean showing at least the minimal clinically important difference (MCID) of 6.4 points).

The secondary endpoint is represented by the safety of the system, which will be assessed by monitoring the frequency and incidence of adverse events. The secondary endpoint evaluation will also assess the overall pain, functional performance, quality of life and radiographic parameters of all enrolled study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 20 years of age or older.
* Patient must be anatomically and structurally suited to receive shoulder arthroplasty implants.
* Patient is a candidate for shoulder arthroplasty due to one or more of the following:

Non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis.

Rheumatoid arthritis. Fractures of the proximal humerus, where other methods of treatment are deemed inadequate.

Difficult clinical management problems, where other method of treatment may not be suitable or may be inadequate.

* Patient must be able and willing to complete the protocol required follow-up.
* Patient must be able and willing to sign the IRB/EC approved informed consent.

Exclusion Criteria:

* Patient is unwilling or unable to give consent or to comply with the follow-up program.
* Patient has any condition which would in the judgement of the Investigator, place the patient at undue risk or interfere with the study.
* Patient is known to be pregnant or breastfeeding.
* Patient is a vulnerable subject (prisoner, mentally incompetent or unable to understand what participation to the study entails, a known alcohol or drug abuser, and/or anticipated to be non- compliant).
* Patient is uncooperative or patient with neurologic disorders who is incapable or unwilling to follow directions.
* Patient has any sign of infection affecting the shoulder joint or in its proximity which may spread to the implant site.
* Patient has rapid joint destruction, marked bone loss, or bone resorption apparent on roentgenogram.
* Patient has any neuromuscular disease compromising the affected limb that would render the procedure unjustifiable.
* Patient presents with osteoporosis, which in the opinion of the Investigator, may limit the subject's ability to support total shoulder arthroplasty using the study device.
* Patient has a metabolic disorder that may impair bone formation.
* Patient has osteomalacia.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Alliance Glenoid is intended to be used as part of an anatomic total shoulder arthroplasty to reduce shoulder pain an improve shoulder function. The Alliance Glenoid is intended to be used as a component of a total shoulder replacement system for primary arthroplasty. It provides the surface on the glenoid side that articulates with the modular head component and stem component on the humeral side. Patients must meet all inclusion and none on the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) | 2 years
  The primary endpoint for this study will be performance assessed by improvement in the American Shoulder and Elbow Surgeons (ASES) shoulder score from baseline to 2 years (as evaluated using the overall cohort mean showing at least the minimal clinically important difference (MCID) of 6.4 points).
  Pain, function, and activities of daily living are measured. The ASES scale is 0-100. 100 is the highest score and indicates the greatest function while 0 is the lowest score.

SECONDARY OUTCOMES:
Frequency and Incidence of Adverse Events (Safety) | 10 years
  Monitoring the frequency and incidence of adverse events, serious adverse events, adverse device effects, serious adverse device effects, and unanticipated serious adverse device effects as well as device deficiencies.
Euroqol Patient Quality of life (EQ-5D-5L) | 10 years
  The EuroQol five dimensions questionnaire (EQ-5D-5L) is a five dimensional self-assessment that is comprised of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. These five dimensions can be used to index a subject's health utility on a scale of 0 to 1, where 0 is death and 1 is perfect health. The scoring rule for EQ-5D permits scores less than 0, implying that some health states may be worse than death.
Radiographic Performance | 10 years
  X-Rays will be evaluated for radiolucency, osteolysis, osteophytes, component migration, subsidence and heterotopic ossification.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Rohmer, Study Director — Zimmer Biomet
Locations (2):
- ARCUS Kliniken Pforzheim, Pforzheim, Germany
- Meander Medisch Centrum, Amersfoort, TZ, Netherlands